CLINICAL TRIAL: NCT03998878
Title: Testing the Effect of Multiple Weight Management Modalities for Chronic Disease Risk Reduction in a Clinical Setting (LIHT)
Brief Title: Testing the Effect of Multiple Weight Management Modalities for Chronic Disease Risk Reduction in a Clinical Setting
Acronym: LIHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1903480167
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Obesity
Keywords: Weight Loss; Diet Modification; Body Weight; Body Weight Changes; Ketogenic diet; Diet, Carbohydrate-Restricted; Fasting; Intermittent Fasting; Hunger training
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight; Body Weight Changes; Fasting; Intermittent Fasting | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Carbohydrate Diet (Experimental): Participants will be instructed to consume less than 30 grams of carbohydrates per day.
  Interventions: Behavioral: Low-Carbohydrate Diet
- Intermittent Energy Restriction (Experimental): Participants choose 2 non-consecutive days per week in which they will consume 500-650 calories.
  Interventions: Behavioral: Intermittent Energy Restriction
- Hunger Training (Experimental): Participants monitor their hunger symptoms and blood glucose, and eat only when blood glucose is below a certain threshold level.
  Interventions: Behavioral: Hunger Training

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diet — Participants will be instructed to follow a low-carbohydrate diet.
  Arms: Low-Carbohydrate Diet
Behavioral: Intermittent Energy Restriction — Participants will be instructed to follow intermittent energy restriction.
  Arms: Intermittent Energy Restriction
Behavioral: Hunger Training — Participants will be instructed to follow Hunger Training.
  Arms: Hunger Training

SUMMARY:
This project will test 3 methods of dietary changes in a weight loss clinic. Participants will be randomized to one of 3 arms: low-carbohydrate diet, intermittent energy restriction, or Hunger Training. A maximum of 30 participants will be assigned to each arm. The goal of the proposed study is to determine the feasibility, early efficacy, and patient satisfaction of each weight loss modality in a population of patients seeking care at a weight loss clinic.

DETAILED DESCRIPTION:
Adult obesity, a common condition in the United States, is a well-established risk factor for the development of chronic diseases, including diabetes, heart disease, hypertension, and many types of cancer. However, research has not determined what type of diet is best for reducing weight and achieving optimal health outcomes. In this randomized trial, participants seeking care at a weight loss clinic will be assigned to one of three diets: low-carbohydrate, intermittent energy restriction, or Hunger Training. On the low-carbohydrate diet, participants will be instructed to consume less than 30 grams of carbohydrates per day. The intermittent energy restriction protocol will require participants to choose 2 non-consecutive days per week in which they will consume 500-650 calories. Hunger Training is a relatively new approach that involves teaching people to monitor their hunger symptoms and blood glucose, and to eat only when blood glucose is below a certain level. To our knowledge, these weight loss modalities have not been compared in a single, clinical study. The goal of the proposed study is to determine the feasibility, early efficacy, and patient satisfaction of each weight loss modality in a population of patients seeking care at a weight loss clinic. The goal will be achieved though the successful completion of the following aims:

Aim 1: To determine the feasibility of recruiting, retaining and maintaining the adherence participants in a randomized clinical trial testing 3 weight loss modalities.

Aim 2: To examine and compare the effect of 3 weight loss modalities on changes in anthropometric measures and metabolic and cancer-related health markers.

Aim 3: To evaluate and compare patients' perceived satisfaction with each weight loss modality.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese as indicated by BMI >27
* Age ≥ 18
* HbA1C <8.0
* Fluent in English

Exclusion Criteria:

* Cognitive state that precludes informed consent or adherence to study protocols
* Pregnant, breast-feeding, or planning to become pregnant within 6 months
* A1C ≥ 8.0
* Taking an anti-obesity medication
* Insulin-dependence
* prior metabolic surgery
* current laparoscopic adjustable gastric band ("lap band") use
* Experience of substantial weight changes (±5 kg or ±10 lbs) in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Rate of Recruitment | 1 year
  Feasibility of recruiting participants into a randomized dietary intervention in a clinic setting as measured by the total number of individuals who are screened as eligible and enrolled into the study
Rate of Retention | 1 year
  Feasibility of retaining participants in a randomized dietary intervention in a clinic setting as measured by the number of participants completing all study visits
Adherence to the Intervention | 1 year
  Feasibility of maintaining participant adherence in a randomized dietary intervention in a clinic setting will be measured by attendance at scheduled clinic visits
Change in Weight | baseline to 3 months
  Participant weight will be measured
Change in BMI | baseline to 3 months
  Participant BMI will be measured
Change in HbA1c | baseline to 3 months
  Participant HbA1c will be measured
Change in Fasting Glucose | baseline to 3 months
  Participant fasting glucose will be measured
Change in Fasting Insulin | baseline to 3 months
  Participant fasting insulin will be measured
Change in Total Cholesterol | baseline to 3 months
  Participant total cholesterol will be measured
Change in Triglycerides | baseline to 3 months
  Participant triglycerides will be measured
Change in High Density Lipoprotein (HDL) | baseline to 3 months
  Participant HDL will be measured
Change in Low Density Lipoprotein (LDL) | baseline to 3 months
  Participant LDL will be measured
Change in C-Reactive Protein (CRP) | baseline to 3 months
  Participant CRP will be measured
Change in Insulin-like Growth Factor 1 (IGF-1) | baseline to 3 months
  Participant IGF-1 will be measured
Change in Insulin-like Growth Factor 2 (IGF-2) | baseline to 3 months
  Participant IGF-2 will be measured
Change in Insulin-like Growth Factor Binding Protein 3 (IGFBP-3) | baseline to 3 months
  Participant IGFBP-3 will be measured
Change in Leptin | baseline to 3 months
  Participant leptin will be measured
Change in Adiponectin | baseline to 3 months
  Participant adiponectin will be measured
Participant Satisfaction | 3 months
  Participants will complete a questionnaire at the end of the study to assess the acceptability of and satisfaction with the weight loss diet intervention they received. We will assess overall satisfaction, enjoyment, likeliness to recommend, and ease of following the diet. Aggregated scores will be compared across weight loss modality.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Algotar, MD, PhD, MPH, Principal Investigator — University of Arizona, Banner University Medical Center; Susan M Schembre, PhD, RD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States